CLINICAL TRIAL: NCT00074282
Title: Phase II Trial of Pentostatin, Cyclophosphamide and Rituximab (PCR) Followed by Campath-1H for Previously Treated Relapsed or Refractory Patients With Chronic Lymphocytic Leukemia
Brief Title: Pentostatin, Cyclophosphamide, and Rituximab Followed By Campath-1H in Patients With Relapsed or Refractory B-Cell CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000343796; E2903 (Other: ECOG-ACRIN)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Pentostatin; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (PCR) (Experimental): Treatment consisted of 6 cycles of pentostatin, cyclophosphamide, and rituximab (PCR) given every 28 days.
  Rituximab administered as follows: For the first infusion, all patients receive 100 mg dose (regardless of weight/BSA). For subsequent infusions, all patients receive rituximab 375 mg/m2.
  Pentostatin and cyclophosphamide administered as follows: Pentostatin given at 4 mg/m2 either as an IV push or IV over 10-30 minutes in 250 mL NS or D5W on day 1 every 4 weeks of cycles 1-6. Cyclophosphamide given at 600 mg/m2 IV over 30-60 minutes in 250 mL NS on day 1 every 4 weeks of cycle 1-6.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: pentostatin
- Arm B (Alemtuzumab: CR, nPR) (Experimental): Patients who achieved a confirmed CR or nPR, were registered to receive Alemtuzumab (Arm B). When the patient was registered to Arm B, the drug was administered three times a week for four weeks. The dose was 30 mg per dose. A twelve-week treatment-free period had to elapse before CAMPATH-1H began following completion of PCR for Arm B patients
  Interventions: Drug: Alemtuzumab
- Arm C (Alemtuzumab: PR, <PR, PD) (Experimental): For those patients not achieving a CR or nPR (thus patients either achieved PR, SD, or PD), Alemtuzumab (Arm C) was administered three times a week for eighteen weeks at a dose of 30 mg TIW. For PR, SD and PD patients, the timing of CAMPATH-1H was left to the discretion of the investigator, and treatment could begin earlier but no less than two weeks and no longer than eight weeks after the completion of the last PCR course. Patients determined to have PD during treatment with PCR did not need to complete all 6 cycles of PCR to go on to Arm C, however, completing a minimum of 2 cycles was required.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
  Arms: Arm A (PCR)
Drug: cyclophosphamide
  Other Names: Cytoxan
  Arms: Arm A (PCR)
Drug: pentostatin
  Other Names: deoxycoformycin; Nipent
  Arms: Arm A (PCR)
Drug: Alemtuzumab
  Other Names: Campath; Campath-1H
  Arms: Arm B (Alemtuzumab: CR, nPR); Arm C (Alemtuzumab: PR, <PR, PD)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pentostatin, cyclophosphamide, and CAMPATH-1H work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well pentostatin, cyclophosphamide, rituximab, and CAMPATH-1H work in treating patients with relapsed or refractory B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate (complete remission, partial remission [PR], or nodular PR) in patients with relapsed or refractory B-cell chronic lymphocytic leukemia (CLL) treated with pentostatin, cyclophosphamide, and rituximab (PCR) followed by CAMPATH-1H .
* Determine the presence of minimal residual disease in patients treated with this regimen who achieve a CR or nPR

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the overall and progression-free survival of patients treated with this regimen.
* Evaluate the number of patients who after PCR (or during PCR for PD), only achieve a PR, SD, or PD and who subsequently convert to a higher response category after CAMPATH-1H .

Exploratory

* Assess the angiogenic profile (i.e., secretion levels of pro- versus anti-angiogenic molecules) of CLL B cell clones as well as bone marrow angiogenesis (i.e., vascular density by immunohistochemistry) at baseline, after PCR, after CAMPATH-1H, every six months (serum only), and at time of response assessment (marrow).
* Determine the V_H gene mutation status and CD38 expression of the B-CLL clones at study entry and at the end of the therapy and assess the association between the VH gene mutation status and CD38 expression and clinical outcome.
* Determine surface phenotype (by flow cytometry) and genetic defects (by CLL FISH panel) information on CLL-B cell clones and associate with clinical outcome.
* Monitor the T-cell status by repertoire and flow cytometry analysis to determine the nature and extent of T-cell deficiency induced by the PCR and CAMPATH-1H treatment and assess any association with clinical outcome and toxicities.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL) meeting the following criteria:

  * Peripheral blood absolute lymphocyte count greater than 5,000/mm^3
  * Lymphocytosis must comprise small to moderate size lymphocytes with no greater than 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
  * Phenotypically characterized CLL defined by the following:

    * Predominant population of cells share B-cell antigens with CD5 in the absence of other pan-T-cell markers (CD3 or CD2)
    * B cell expresses either kappa or lambda light chains
    * Surface immunoglobulin with low cell surface density expression
* Requires chemotherapy, as indicated by any of the following:

  * Disease-related symptoms

    * Weight loss of 10% or more within the past 6 months
    * Extreme fatigue
    * Fevers greater than 100.5°F for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure manifested by the development of or worsening anemia (hemoglobin no greater than 10 g/dL) and/or thrombocytopenia (platelet count no greater than 100,000/mm^3)
  * Massive (i.e., greater than 6 cm below left costal margin) or progressive splenomegaly
  * Massive nodes or clusters (i.e., greater than 10 cm in longest diameter) or progressive adenopathy
  * Progressive lymphocytosis with an increase of greater than 50% over a 2-month period OR an anticipated doubling time of less than 6 months
* Demonstrated progression after at least 1 course of either an alkylating agent-based or purine nucleoside-based (e.g., fludarabine) regimen OR failed to achieve a meaningful response OR relapsed after prior therapy

  * Patients who have relapsed after a pentostatin-based regimen are eligible provided the response was greater than 12 months prior to study entry
* 18 and over
* ECOG Performance Status 0-2
* Bilirubin no greater than 2 mg/dL (unless secondary to tumor, hemolysis, or Gilbert syndrome)
* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance ≥ 30 mL/min
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception (including 1 barrier method) for at least 28 days before starting lenalidomide, while participating in the study, and for at least 28 days after discontinuation/stopping lenalidomide
* At least 8 weeks since prior rituximab
* At least 6 weeks since prior chemotherapy
* At least 1 year since prior pentostatin, cyclophosphamide, and rituximab (PCR) therapy

  * PCR therapy at least 1 year prior to study entry allowed

Exclusion criteria:

* Bone marrow dysplasia related to prior therapy
* New York Heart Association class III or IV heart failure
* Prior lenalidomide
* Other malignancy within the past 2 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* Pregnant or nursing
* Concurrent oral or IV antibiotics for active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-04-14 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2018-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanford J. Kempin, MD, Study Chair — Beth Israel Medical Center
Locations (143):
- United States (143):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - New Orleans Cancer Institute at Memorial Medical Center, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Union Hospital of Cecil County, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Kay NE, Kim HT, Kempin S, et al.: Predictors of clinical outcome to pentostatin, cyclophosphamide and rituximab (PCR) followed by campath for relapsed/refractory CLL : a study of the Eastern Cooperative Oncology Group, E2903. [Abstract] Blood 112 (11): A-1057, 2008.
- [Result] Kempin S, Kay NE, Sun Z, et al.: Early results of pentostatin, cytoxan, rituximab (PCR) followed by CAMPATH-H (CA) for the treatment of relapse/refractory chronic lymphocytic leukemia (CLL) in ECOG protocol E2903. [Abstract] Blood 110 (11): A-3109, 2007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from ECOG-ACRIN institutions between 12/16/04 and 5/6/13. The first patient was accrued on 4/14/05.
Groups:
- Arm A (PCR): Treatment consisted of 6 cycles of pentostatin, cyclophosphamide, and rituximab (PCR) given every 28 days.
  Rituximab administered as follows: For the first infusion, all patients receive 100 mg dose (regardless of weight/BSA). For subsequent infusions, all patients receive rituximab 375 mg/m2.
  Pentostatin and cyclophosphamide administered as follows: Pentostatin given at 4 mg/m2 either as an IV push or IV over 10-30 minutes in 250 mL NS or D5W on day 1 every 4 weeks of cycles 1-6. Cyclophosphamide given at 600 mg/m2 IV over 30-60 minutes in 250 mL NS on day 1 every 4 weeks of cycle 1-6.
  rituximab
  cyclophosphamide
  pentostatin
- Arm B (Alemtuzumab: CR, nPR): Patients who achieved a confirmed CR or nPR, were registered to receive Alemtuzumab (Arm B). When the patient was registered to Arm B, the drug was administered three times a week for four weeks. The dose was 30 mg per dose. A twelve-week treatment-free period had to elapse before CAMPATH-1H began following completion of PCR for Arm B patients
  Alemtuzumab
- Arm C (Alemtuzumab: PR, <PR, PD): For those patients not achieving a CR or nPR (thus patients either achieved PR, SD, or PD), Alemtuzumab (Arm C) was administered three times a week for eighteen weeks at a dose of 30 mg TIW. For PR, SD and PD patients, the timing of CAMPATH-1H was left to the discretion of the investigator, and treatment could begin earlier but no less than two weeks and no longer than eight weeks after the completion of the last PCR course. Patients determined to have PD during treatment with PCR did not need to complete all 6 cycles of PCR to go on to Arm C, however, completing a minimum of 2 cycles was required.
  Alemtuzumab
Period: Step 1
Arm/Group | Arm A (PCR) | Arm B (Alemtuzumab: CR, nPR) | Arm C (Alemtuzumab: PR, <PR, PD)
Started | 102 | 0 | 0
Eligible | 98 | 0 | 0
Started Treatment | 96 | 0 | 0
Completed | 44 | 0 | 0
Not Completed | 58 | 0 | 0
Not completed — Adverse Event | 32 | 0 | 0
Not completed — Death | 6 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0
Not completed — Disease progression | 2 | 0 | 0
Not completed — Alternative therapy | 2 | 0 | 0
Not completed — Other complicating disease | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Ineligible | 4 | 0 | 0
Not completed — Never started treatment | 2 | 0 | 0
Period: Step 2
Arm/Group | Arm A (PCR) | Arm B (Alemtuzumab: CR, nPR) | Arm C (Alemtuzumab: PR, <PR, PD)
Started | 0 | 9 | 31
Completed | 0 | 7 | 7
Not Completed | 0 | 2 | 24
Not completed — Adverse Event | 0 | 2 | 12
Not completed — Disease progression | 0 | 0 | 5
Not completed — Death | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who began treatment
Arm/Group | Arm A (PCR)
Number analyzed (Participants) | 96
Age, Continuous [Median (Full Range); unit: years] | 64 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 92
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percent with response (CR, nPR, PR) with two-stage 90% confidence interval
Time Frame: 8 weeks after Cycle 6
Population: Eligible patients who began treatment
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Arm A (PCR)
Number analyzed (Participants) | 96
percentage | 55.2 [46.3 to 63.9]

2. Primary Outcome: Molecular Complete Remission (MCR) Rate
Description: Percent of patients who have MCR (clinical CR with flow negative and RT-PCR negative)
Time Frame: 3 months post alemtuzumab
Population: Patients who achieved a CR or nPR in Step 1 and were eligible for and began treatment on Step 2
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | Arm B (Alemtuzumab: CR, nPR)
Number analyzed (Participants) | 9
percentage | 44.4 [16.9 to 74.9]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from registration until death from any cause.
Time Frame: Up to 5 years from registration
Population: Eligible patients who began treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (PCR)
Number analyzed (Participants) | 96
months | 27.6 [20.2 to 42.2]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from registration until induction failure, institution of non-protocol therapy, relapse or death from any cause in the absence of relapse.
Time Frame: Up to 5 years from registration
Population: Eligible patients who began treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (PCR)
Number analyzed (Participants) | 96
months | 12.2 [9.7 to 14.5]

5. Secondary Outcome: Number of Patients Who After PCR (or During PCR for PD), Only Achieve a PR, SD, or PD and Who Subsequently Convert to a Higher Response Category After Campath-1H
Time Frame: From re-registration up to 5 years (followed for response until progression)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm C (Alemtuzumab: PR, <PR, PD)
Number analyzed (Participants) | 30
Participants | 4

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (PCR) | Arm B (Alemtuzumab: CR, nPR) | Arm C (Alemtuzumab: PR, <PR, PD)
All-Cause Mortality (participants affected / at risk) | 71/100 | 5/9 | 23/31
Serious Adverse Events (participants affected / at risk) | 88/100 | 8/9 | 31/31
Other Adverse Events (participants affected / at risk) | 99/100 | 9/9 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (PCR) (N=100) | Arm B (Alemtuzumab: CR, nPR) (N=9) | Arm C (Alemtuzumab: PR, <PR, PD) (N=31)
Allergic reaction (Immune system disorders) | 3 | 0 | 0
CD4 decreased (Investigations) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 16 | 1 | 7
Leukocytes decreased (Investigations) | 1 | 1 | 2
Lymphopenia (Investigations) | 38 | 8 | 28
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Neutrophils decreased (Investigations) | 60 | 4 | 17
Platelets decreased (Investigations) | 34 | 3 | 13
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac-ischemia (Cardiac disorders) | 1 | 0 | 0
C-P arrest, non-fatal, cause unknown (Cardiac disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1
Fatigue (General disorders) | 9 | 0 | 4
Fever w/o neutropenia (General disorders) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1
Death - multiorgan failure (General disorders) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 1 | 5
Infection w/ gr3-4 neut, lung (Infections and infestations) | 3 | 0 | 4
Infection w/ gr3-4 neut, sinus (Infections and infestations) | 0 | 0 | 2
Infection w/ gr3-4 neut, skin (Infections and infestations) | 2 | 0 | 1
Infection Gr0-2 neut, catheter (Infections and infestations) | 1 | 0 | 0
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 0 | 0 | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 4 | 0 | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 2 | 0 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 1 | 0 | 1
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 1 | 0
Infection-other (Infections and infestations) | 0 | 0 | 0
Edema limb (General disorders) | 2 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Creatinine increased (Investigations) | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 1 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Speech impairment (Nervous system disorders) | 1 | 0 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest/thoracic pain NOS (General disorders) | 1 | 0 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neuropathic, pain (Nervous system disorders) | 1 | 0 | 0
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cystitis (Renal and urinary disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 6 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 0 | 0
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 6 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (PCR) (N=100) | Arm B (Alemtuzumab: CR, nPR) (N=9) | Arm C (Alemtuzumab: PR, <PR, PD) (N=31)
Allergic reaction (Immune system disorders) | 18 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 93 | 8 | 30
Lymphopenia (Investigations) | 58 | 2 | 14
Neutrophils decreased (Investigations) | 56 | 5 | 23
Platelets decreased (Investigations) | 74 | 7 | 24
Hypertension (Vascular disorders) | 6 | 0 | 2
Hypotension (Vascular disorders) | 7 | 0 | 0
Fatigue (General disorders) | 72 | 5 | 21
Fever w/o neutropenia (General disorders) | 26 | 3 | 6
Insomnia (Psychiatric disorders) | 15 | 1 | 0
Rigors/chills (General disorders) | 31 | 4 | 9
Sweating (Skin and subcutaneous tissue disorders) | 10 | 2 | 5
Weight loss (Investigations) | 20 | 2 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Injection site reaction (General disorders) | 0 | 2 | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hot flashes (Vascular disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 25 | 3 | 6
Constipation (Gastrointestinal disorders) | 16 | 1 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 24 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 11 | 0 | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 10 | 0 | 4
Nausea (Gastrointestinal disorders) | 66 | 2 | 10
Taste disturbance (Nervous system disorders) | 14 | 2 | 3
Vomiting (Gastrointestinal disorders) | 39 | 1 | 5
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 0 | 0 | 2
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 0 | 1 | 0
Edema limb (General disorders) | 15 | 0 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 21 | 3 | 9
Aspartate aminotransferase increased (Investigations) | 31 | 2 | 6
Acidosis (Metabolism and nutrition disorders) | 14 | 2 | 1
Blood bilirubin increased (Investigations) | 19 | 1 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 41 | 3 | 10
Creatinine increased (Investigations) | 29 | 1 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 61 | 5 | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 15 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 12 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 7 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 28 | 2 | 8
Hyperuricemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 8 | 2 | 3
Depression (Psychiatric disorders) | 0 | 1 | 6
Neuropathy-motor (Nervous system disorders) | 0 | 1 | 1
Neuropathy-sensory (Nervous system disorders) | 12 | 1 | 4
Ocular-other (Eye disorders) | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 7 | 1 | 2
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Head/headache (Nervous system disorders) | 14 | 1 | 4
Joint, pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 15 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 2 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 3 | 8
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cystitis (Renal and urinary disorders) | 5 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT00074282/Prot_SAP_000.pdf